CLINICAL TRIAL: NCT00084409
Title: A Randomized Phase II Chemoprevention Study of Iloprost Versus Placebo in Patients at High Risk for Lung Cancer
Brief Title: Iloprost in Preventing Lung Cancer in Patients at High Risk for This Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-279.cc; National Cancer Institute (Other Grant/Funding Number: P50CA058187); 01-279 (Other: IRB Number from OnCore)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; squamous lung dysplasia
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral iloprost twice daily for 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: iloprost
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily for 6 months in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: iloprost — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Iloprost may be effective in preventing lung cancer.

PURPOSE: This randomized phase II trial is studying how well iloprost works in preventing lung cancer in patients who are at high risk for this disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the reversal of premalignant histological changes in the bronchial epithelium of patients at high risk for lung cancer (defined by > 20 pack years of smoking and sputum atypia) treated with iloprost vs placebo.
* Determine whether this drug modulates Ki-67 proliferation index (Antigen Ki-67) in these patients.
* Determine whether this drug affects prostaglandin metabolism in these patients.
* Determine the toxicity profile of this drug in these patients.

Secondary

* Determine whether this drug modulates a panel of biomarkers, including MCM-2(Minichromosome maintenance protein: forms DNA helicase), EGFR (Epidermal growth factor receptor: cell surface receptor for the epidermal growth factor family of proteins. Mutations in EGFR expression or activity can result in cancer.) , HER2/neu (Human epidermal growth factor receptor 2 HER2 is a member of the EGFR family), RARβ (Retinoic Acic Receptor Beta is a nuclear transcription regulator and a member of the thyroid-steroid hormone receptor superfamily), p53, FHIT (Fragile histidine triad protein is an enzyme involved in purine metabolism and had been demonstrated to be a tumor suppressor), apoptotic index, and microvessel density, in these patients.
* Determine the genes whose expression is altered by this drug in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to smoking status (current vs former) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral iloprost twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 6 months in the absence of unacceptable toxicity.

Patients are followed at 1 month and then annually thereafter.

PROJECTED ACCRUAL: A total of 152 patients (76 [38 current smokers and 38 former smokers] per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smoker with ≥ 20 pack-year history of smoking with no tobacco use within the past 6 months
* Mild atypia or worse on sputum cytology, or
* Bronchial biopsy with mild or worse dysplasia within the past 12 months
* Age 18 and over
* SWOG (Southwest Oncology Group)0-2
* Life expectancy at least 6 months
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* Transaminases ≤ 2.5 times ULN
* Bilirubin ≤ 2.0 mg/dL
* Albumin ≥ 2.5 g/dL
* Creatinine ≤ 1.5 mg/dL
* Well-controlled atrial fibrillation OR rare (< 2 minutes) premature ventricular contractions allowed
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able and willing to undergo bronchoscopy

Exclusion Criteria

* Clinically apparent bleeding diathesis
* Ventricular tachycardia
* Multifocal premature ventricular contractions or supraventricular tachycardias with rapid ventricular response
* Pneumonia or acute bronchitis within the past 2 weeks
* Hypoxemia (< 90% saturation with supplemental oxygen)
* Pregnant or nursing
* Malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Serious medical condition that would preclude bronchoscopy or study participation
* Clinically active coronary artery disease
* Myocardial infarction within the past 6 weeks
* Chest pain
* Congestive heart failure
* Cardiac dysrhythmia that is potentially life-threatening

Exclusion for PRIOR CONCURRENT THERAPY:

* Biologic therapy (Not specified)
* More than 5 years since prior chemotherapy
* More than 6 weeks since prior inhaled steroids
* More than 5 years since prior thoracic radiotherapy
* Surgery (Not specified)
* No prior prostacyclin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2001-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Keith, MD, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Keith RL, Blatchford PJ, Kittelson J, Minna JD, Kelly K, Massion PP, Franklin WA, Mao J, Wilson DO, Merrick DT, Hirsch FR, Kennedy TC, Bunn PA Jr, Geraci MW, Miller YE. Oral iloprost improves endobronchial dysplasia in former smokers. Cancer Prev Res (Phila). 2011 Jun;4(6):793-802. doi: 10.1158/1940-6207.CAPR-11-0057. PMID 21636546
- See also: ClinicalTrials.Gov — https://clinicaltrials.gov/ct2/show/NCT00084409?cond=Iloprost&draw=4&rank=32

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The majority of patients were recruited between November 2002 and July 2008 from from pulmonary medicine clinics.
Pre-assignment Details: Patients were excluded from randomization according to the exclusion criteria which included prior history of cancer, significant comorbid disease or inability to undergo 2 bronchoscopies, hypoxemia with the required use of supplemental oxygen, use of inhaled steroids within 6 weeks of enrollment, and carcinoma in situ or invasive cancer on bronch.
Groups:
- Iloprost: Patients receive oral iloprost twice daily for 6 months in the absence of unacceptable toxicity.This group consisted of current and former smokers.
- Placebo: Patients receive oral placebo twice daily for 6 months in the absence of unacceptable toxicity.This group consisted of current and former smokers.
Period: Overall Study
Arm/Group | Iloprost | Placebo
Started | 75 (40 Current, 35 former) | 77 (41 current, 36 former)
Completed | 60 (9 current, 6 former) | 65 (4 Current, 8 former)
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloprost | Placebo | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 62 | 119
  >=65 years | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11) | 58 (9) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 52 | 58 | 110
Region of Enrollment [Number; unit: participants]
  United States | 75 | 77 | 152

OUTCOME MEASURES:

1. Primary Outcome: Change in Average (Follow-up - Baseline) From All Biopsies
Description: This outcome measure is created for each subject as follows:
  From all biopsies scored at the baseline bronchoscopy, the mean WHO score is calculated.
  From all biopsies scored at the follow-up bronchoscopy, the mean WHO score is calculated.Histology on bronchial biopsies pre-treatment and post-treatment will be compared. All biopsies will be graded according to the WHO classification for bronchial epithelium for this outcome, and all the following outcomes.
  WHO Classification Grade Normal 1.0 Reserve Cell Hyperplasia 2.0 Metaplasia 3.0 Mild Dysplasia 4.0 Moderate Dysplasia 5.0 Severe Dysplasia 6.0 Carcinoma in Situ 7.0 Carcinoma 8.0
  The difference (follow-up mean - baseline mean) is used as the outcome measure for each subject.
Time Frame: Nine years
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
WHO Units | -0.23 (0.77) | -0.02 (0.79)

2. Secondary Outcome: Change in Dysplasia Index (Follow-up - Baseline) Using All Biopsies
Description: This outcome measure is created for each subject as follows:
  From all biopsies scored at the baseline bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated (this is the definition of Dysplasia Index (DI)).
  From all biopsies scored at the follow-up bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated.
  The difference (follow-up DI - baseline DI) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: Percentage points
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
Percentage points | -7.70 (21.76) | -0.92 (25.23)

3. Secondary Outcome: Change in Average (Follow-up - Baseline) Using Reference Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are those from the following 6 anatomical sites pre-specified in the protocol to be biopsied: RUL (Right upper lobe: the superior region of the right lung), RML (Right middle lobe: an anatomic portion of the right lung), RB6 (The carina in the right lower lobe at the entrance to the superior segment), LUL (Left upper lobe: the superior portion of the lung), LUDB (Left upper division bronchus: the carina between the lingular orifice and the left upper lobe), and LB6 (The carina in the left lower lobe at the entrance to the superior segment).
  From these biopsies scored at the baseline bronchoscopy, the mean WHO score is calculated.
  From these biopsies scored at the follow-up bronchoscopy, the mean WHO score is calculated.
  The difference (follow-up mean - baseline mean) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
WHO Units | -0.23 (0.82) | -0.01 (0.82)

4. Secondary Outcome: Change in Maximum (Follow-up - Baseline) Using Reference Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are those from the following 6 anatomical sites pre-specified in the protocol to be biopsied: RUL, RML, RB6, LUL, LUDB, and LB6.
  From these biopsies scored at the baseline bronchoscopy, the maximum WHO score is used.
  From these biopsies scored at the follow-up bronchoscopy, the maximum WHO score is used.
  The difference (follow-up maximum - baseline maximum) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
WHO Units | -0.35 (1.58) | 0.11 (1.30)

5. Secondary Outcome: Change in Dysplasia Index (Follow-up - Baseline) Using Reference Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are those from the following 6 anatomical sites pre-specified in the protocol to be biopsied: RUL, RML, RB6, LUL, LUDB, and LB6.
  From these biopsies scored at the baseline bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated (this is the definition of Dysplasia Index (DI)).
  From these biopsies scored at the follow-up bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated.
  The difference (follow-up DI - baseline DI) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: Percentage points
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
Percentage points | -7.61 (23.43) | 0.15 (26.41)

6. Secondary Outcome: Change in Average (Follow-up - Baseline) Using Matched Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies, thus creating "pairs" of biopsies.
  From these biopsies scored at the baseline bronchoscopy, the mean WHO score is calculated.
  From these biopsies scored at the follow-up bronchoscopy, the mean WHO score is calculated.
  The difference (follow-up mean - baseline mean) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
WHO Units | -0.24 (0.78) | -0.06 (0.86)

7. Secondary Outcome: Change in Maximum (Follow-up - Baseline) Using Matched Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies.
  From these biopsies scored at the baseline bronchoscopy, the maximum WHO score is used.
  From these biopsies scored at the follow-up bronchoscopy, the maximum WHO score is used.
  The difference (follow-up maximum - baseline maximum) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
WHO Units | -0.53 (1.46) | 0.11 (1.26)

8. Secondary Outcome: Change in Dysplasia Index (Follow-up - Baseline) Using Matched Sites
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies.
  From these biopsies scored at the baseline bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated (this is the definition of Dysplasia Index (DI)).
  From these biopsies scored at the follow-up bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated.
  The difference (follow-up DI - baseline DI) is used as the outcome measure for each subject.
Time Frame: 9 Years
Measure: Mean (Standard Deviation); unit: Percentage points
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 60 | 65
Percentage points | -7.97 (22.13) | -2.34 (25.49)

9. Secondary Outcome: Change in Average (Follow-up - Baseline) Using Baseline Non-Normal Pairs
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies, thus creating "pairs" of biopsies. Any "pair" for which the baseline WHO score was 1 (i.e. normal tissue) was excluded from the analysis.
  From these biopsies scored at the baseline bronchoscopy, the mean WHO score is calculated.
  From these biopsies scored at the follow-up bronchoscopy, the mean WHO score is calculated.
  The difference (follow-up mean - baseline mean) is used as the outcome measure for each subject.
Time Frame: 9 Years
Population: The analysis was restricted to the 107 subjects (52 in the iloprost group, 55 in the placebo group) with at least 1 non-normal biopsy at baseline, thereby excluding the 18 subjects (8 in the iloprost group and 10 in the placebo group) who had only normal biopsy tissue at baseline.
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 52 | 55
WHO Units | -0.71 (0.93) | -0.38 (0.99)

10. Secondary Outcome: Change in Maximum (Follow-up - Baseline) Using Baseline Non-Normal Pairs
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies, thus creating "pairs" of biopsies. Any "pair" for which the baseline WHO score was 1 (i.e. normal tissue) was excluded from the analysis.
  From these biopsies scored at the baseline bronchoscopy, the maximum WHO score is used.
  From these biopsies scored at the follow-up bronchoscopy, the maximum WHO score is used.
  The difference (follow-up maximum - baseline maximum) is used as the outcome measure for each subject.
Time Frame: 9 Years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: WHO Units
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 52 | 55
WHO Units | -0.81 (1.46) | -0.13 (1.26)

11. Secondary Outcome: Change in Dysplasia Index (Follow-up - Baseline) Using Baseline Non-Normal Pairs
Description: This outcome measure is created for each subject as follows:
  The biopsies used in this analysis are restricted to biopsies from anatomical sites that were biopsies during both the baseline and follow-up bronchoscopies, thus creating "pairs" of biopsies. Any "pair" for which the baseline WHO score was 1 (i.e. normal tissue) was excluded from the analysis.
  From these biopsies scored at the baseline bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated (this is the definition of Dysplasia Index (DI)).
  From these biopsies scored at the follow-up bronchoscopy, the percentage with a WHO score greater than or equal to 4 is calculated.
  The difference (follow-up DI - baseline DI) is used as the outcome measure for each subject.
Time Frame: 9 Years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage points
Arm/Group | Iloprost | Placebo
Number analyzed (Participants) | 52 | 55
Percentage points | -14.32 (31.39) | -6.48 (34.26)

12. Other Pre Specified Outcome: To Determine if Iloprost Can Modulate K-67 Proliferation Index in Patients at High Risk to Develop Lung Cancer
Time Frame: nine years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: To Determine Whether Iloprost Affects Prostaglandin Metabolism by Examining 4 Markers, PGIS, COX-2, PPAR and PPAR.
Description: PGIS (Prostacyclin synthase: an enzyme in the eicosanoid pathway that catalyzes the conversion of prostaglandin H2 to prostaglandin I2 (prostacyclin). PPAR (Peroxisome proliferator-activated receptor: a group of nuclear receptor proteins that act as transcription factors regulating gene expression),
Time Frame: Nine years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: To Determine the Toxicity Profile of Iloprost in Patients at High Risk to Develop Lung Cancer.
Time Frame: Nine Years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Define the Genes Whose Expression is Altered by Iloprost Treatment by Gene Expression Arrays and Quantitative PCR.
Time Frame: Nine Years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: To Determine Whether Iloprost Can Modulate a Panel of Biomarkes.
Description: To determine if Iloprost can modulate a panel of biomarkers including MCM-2, EGFR, Her-2/neu, RARβ, p53, FHIT, apoptotic index, and microvessel density.
Time Frame: 9 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 Years
Description: Adverse event collection was obtained at monthly visits on all randomized participants according to the NCI CommonToxicity criteria version 2.0, entered in case report forms, and in the NCI Oracle Clinical Database
Arm/Group | Iloprost | Placebo
Serious Adverse Events (participants affected / at risk) | 3/75 | 6/77
Other Adverse Events (participants affected / at risk) | 52/75 | 32/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost (N=75) | Placebo (N=77)
Hospitalization (General disorders) | 3 | 4 — SAE(Serious Adverse Event) was reported on subjects who were hospitalized. None of these subjects had > Grade 3 toxicities reported, and the hospitalizations were not attributed to either the drug or placebo.
Death (General disorders) | 0 | 1 — Subject's death was reported as an SAE. The death was not attributed to being on the clinical trial. The subject was on a placebo
CVA - Stroke (Nervous system disorders) | 0 | 1 — Patient suffered a stroke. Patient was on the Placebo
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost (N=75) | Placebo (N=77)
Headache (Nervous system disorders) | 40 | 17
Flushing (Vascular disorders) | 18 | 6
Nausea (Gastrointestinal disorders) | 12 | 6
Pain - Other (General disorders) | 12 | 6
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 13 | 1
Fatigue (General disorders) | 8 | 2
Metabolic/Laboratory - Other (Investigations) | 3 | 6
Neuropathic pain (Nervous system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes